CLINICAL TRIAL: NCT01334892
Title: A Phase II, Multicentre, Randomised, Double-blind, Placebo Controlled Clinical Trial to Investigate the Efficacy and Safety of Aerosolised Liposomal Ciclosporin A Versus Aerosolised Placebo in the Prevention of Bronchiolitis Obliterans Syndrome in Lung Transplant Patients
Brief Title: L-CsA in the Prevention of Bronchiolitis Obliterans Syndrome (BOS) in Lung Transplant (LT) Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim analysis results revealed substantial increase of patient number, with unfeasible study prolongation.
Sponsor: Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12011.201; 2008-003800-73 (EudraCT Number); ISRCTN66069132 (Registry Identifier: ISRCTN66069132)
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-CsA (Active Comparator): Twice daily inhalation of 2.5 ml/10 mg L-CsA for 96 weeks
  Interventions: Drug: Cyclosporine Inhalation Solution
- L-CsA placebo (Placebo Comparator): Twice daily inhalation of 2.5 ml aerosolised placebo (carrier) for 96 weeks (24 months)
  Interventions: Drug: Cyclosporine Inhalation Solution

INTERVENTIONS:
Drug: Cyclosporine Inhalation Solution — Cyclosporin for inhalation twice daily

SUMMARY:
Immunosuppression is a key intervention in patients with solid organ transplant and is usually achieved by combination therapy with systemic CsA or tacrolimus with azathioprine, mycophenolate mofetil (MMF), or corticoids. However, the outcomes after lung transplantation are poor when compared with those after heart, kidney, or liver transplantation, with a survival rate of only 55% for recipients of lung transplants.

Additional application of aerosolised L-CsA should suppress T-cell activation in the lung tissue and subsequently BOS development. The overall purpose of this phase-II/III study is to obtain efficacy and safety data of L-CsA in the prevention of BOS.

DETAILED DESCRIPTION:
Preventive therapeutic intervention by L-CsA is primarily aimed to suppress T-lymphocyte suppression and inflammatory responses and secondly to prevent fibrotic effects making it more likely to be effective in early stages of BOS. Early development of BOS, which mostly will not be diagnosed, and acute organ rejections are strongly patho-physiological associated. Prevention of the very early development of chronic rejection by L-CsA post LTX may be the ideal starting point for IMP application.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent
2. Received a single lung, bilateral lung or heart/lung transplantation between 6 weeks and 26 weeks prior to first IMP administration.
3. Male or female, 18 years of age
4. Capable of self-administration of medications
5. Capable of understanding the purpose and risk of the clinical trial
6. Received the following immunosuppressive agents and dosages for maintenance therapy:

   1. Tacrolimus and
   2. Mycophenolate mofetil (MMF) 1 to 3 g/day and
   3. Prednisone or any other steroid therapy; tapered down
7. Female patients with childbearing potential must have a negative urine pregnancy test prior to first IMP administration.
8. Estimated life expectancy > 6 month

Exclusion Criteria:

1. Any previous episode of bronchiolitis obliterans (BO) or bronchiolitis obliterans syndrome (BOS) of grade 1 or higher
2. Any active invasive bacterial, viral or fungal infection
3. Received systemic maintenance immunosuppressive therapy other than listed in the inclusion criteria
4. Received any systemic or topical ciclosporin A within
5. Received any systemic or topical Rosuvastatin
6. Current mechanical ventilation
7. Received a lung re-transplantation
8. Pregnant or breast feeding woman
9. Has known hypersensitivity to ciclosporin A
10. Has a serum creatinine value of more than 265 µmol/L (3 mg/dL)
11. Unlikely to comply with visits, inhalation procedures or spirometric measurements
12. Receipt of an investigational drug within 4 weeks prior to first administration of IMP
13. Any co-existing medical condition that in the investigator's judgement
14. Psychiatric disorders or altered mental status
15. Patient was previously enrolled in the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare cumulative BOS-free survival of patients recieving L-CsA or placebo. | 2 years
  BOS stage 1 and higher is considered as BOS for the primary endpoint.

SECONDARY OUTCOMES:
Cumulative mean incidence of BOS 12, 18 and 24 months after first IMP administration | 2 years
  Further secondary objectives are to compare further efficacy and safety data from L-CsA versus placebo. Evaluation of IMP pharmacokinetic (PK) data in whole blood samples and bronchoalveolar lavage (BAL)are included in the outcome measure.
  The main safety evaluation is the incidence of treatment-emergent AEs including clinically relevant laboratory parameters and vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- PARI Pharma GmbH, Gräfelfing, Germany